CLINICAL TRIAL: NCT04724239
Title: A Randomized Phase 2 Clinical Trial Evaluating Sintilimab and Chidamide in Combination With or Without IBI305 in Patients With Standard Treatment Failure of Advanced or Metastatic pMMR/MSS Colorectal Carcinoma
Brief Title: Sintilimab and Chidamide in Combination With or Without IBI305 in Advanced or Metastatic pMMR/MSS Colorectal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, The president of Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPability-01
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Advanced Microsatellite Stable Colorectal Cancer; Metastatic Microsatellite-stable Colorectal Cancer
Keywords: Colorectal Carcinoma, pMMR, Microsatellite-stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in approximately a 1:1 ratio to receive sintilimab and chidamide with or without IBI305.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The triplet group (sintilimab + chidamide + IBI305) (Experimental): Every 3 weeks, patients received sintilimab 200 mg and IBI305(bevacizumab) 7.5 mg/kg on day one and chidamide 30 mg orally twice weekly.
  Interventions: Drug: Sintilimab; Drug: Chidamide; Drug: IBI305
- The doublet group (sintilimab + chidamide) (Active Comparator): Every 3 weeks, patients received sintilimab 200 mg on day one and chidamide 30 mg orally twice weekly.
  Interventions: Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Sintilimab — 200mg IV on Day 1 Q3W
Drug: Chidamide — 30mg PO BIW each 3-week cycle
Drug: IBI305 — 7.5mg/kg IV on Day 1 Q3W
  Other Names: Bevacizumab
  Arms: The triplet group (sintilimab + chidamide + IBI305)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sintilimab and chidamide in combination with or without IBI305(bevacizumab) in patients with standard treatment failure of advanced or metastatic pMMR/MSS colorectal adenocarcinoma.

DETAILED DESCRIPTION:
In this study, we explored the potential effectiveness of combining PD-1 monoclonal antibody sintilimab with the histone deacetylase inhibitor (HDACi) chidamide, with or without IBI305(bevacizumab), in MSS/pMMR unresectable locally advanced or metastatic colorectal cancer patients who failed standard chemotherapy and testified this new combination in preclinical models. Fourty-eight patients were randomized into two groups: the doublet group, who received sintilimab 200 mg every 3 weeks and chidamide 30 mg orally twice weekly, and the triplet group, who received sintilimab, chidamide, and bevacizumab 7.5 mg/kg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of unresectable locally advanced, recurrent or metastatic colorectal adenocarcinoma.
2. Tumor tissues were identified as mismatch repair-proficient (pMMR) by immunohistochemistry (IHC) method or microsatellite stability (MSS) by polymerase chain reaction (PCR).
3. Subjects must have failed at least two lines of prior treatment.
4. Subjects must have one measurable lesion according to RECIST v1.1 at least.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. 18-75 years old.
7. Life expectancy of at least 12 weeks.
8. Adequate bone marrow, liver, renal and coagulation function as assessed by the laboratory required by protocol

Exclusion Criteria:

1. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody or histone deacetylase (HDAC) inhibitor.
2. Received last dose of anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy or arterial embolization) within 3 weeks of the first dose of study medication.
3. Received radiotherapy with 4 weeks of the first dose of study medication.
4. Underwent major operation within 4 weeks of the first dose of study medication or open wound, ulcer or fracture.
5. Known symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Subjects received prior treatment and have stable disease more than 4 weeks from first dose of study medication are permitted to enroll.
6. Active, known or suspected autoimmune disease or has a history of the disease within the last 2 years.
7. Interstitial lung disease requiring corticosteroids.
8. Active or poorly controlled serious infections.
9. Significant malnutrition.
10. Symptomatic congestive heart failure (NYHA Class II-IV) or symptomatic or poorly controlled arrhythmia.
11. Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment.
12. Within 6 months prior to the enrollment, history of gastrointestinal perforation and/or fistula, gastrointestinal ulcer, bowel obstruction, extensive bowel resection, Crohn's disease, or ulcerative colitis, intra-abdominal abscesses, or long-term chronic diarrhea.
13. History or evidence of inherited bleeding diathesis or coagulopathy or thrombus
14. Any life-threatening bleeding within 3 months prior to the enrollment.
15. High risk of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival (PFS) rates at 18 weeks | 24 months
  The proportion of patients without disease progression or death at the 18th week after initiation of the study treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 year
  The proportion of patients with a PR or CR
Progression-free survival (PFS); | 2 year
  The time from enrollment until tumor progression or death from any cause, whichever occurred first
Overall Survival (OS); | 2 year
  The time calculated from enrollment until death from any cause, with living patients censored at the last known survival date
Disease control rate (DCR) | 2 year
  The proportion of patients with a PR, CR, or SD
Duration of response (DoR) | 2 year
  For patients who achieved a complete response (CR) or partial response (PR), the time from the first tumor assessment demonstrating response until disease progression or death, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang F, Jin Y, Wang M, Luo HY, Fang WJ, Wang YN, Chen YX, Huang RJ, Guan WL, Li JB, Li YH, Wang FH, Hu XH, Zhang YQ, Qiu MZ, Liu LL, Wang ZX, Ren C, Wang DS, Zhang DS, Wang ZQ, Liao WT, Tian L, Zhao Q, Xu RH. Combined anti-PD-1, HDAC inhibitor and anti-VEGF for MSS/pMMR colorectal cancer: a randomized phase 2 trial. Nat Med. 2024 Apr;30(4):1035-1043. doi: 10.1038/s41591-024-02813-1. Epub 2024 Mar 4. PMID 38438735